CLINICAL TRIAL: NCT05497089
Title: Temelimab as a Disease Modifying Therapy in Patients With Neurological, Neuropsychological, and Psychiatric (=Neuropsychiatric) Symptoms in Post-COVID 19 or Postacute Sequelae of COVID-19 (PASC) Syndrome
Brief Title: Temelimab as a Disease Modifying Therapy in Patients With Neuropsychiatric Symptoms in Post-COVID 19 or PASC Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GeNeuro SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-501; 2022-000618-32 (EudraCT Number)
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Post-COVID-19 Syndrome
Keywords: GNbAC1; Human Endogenous Retrovirus Type W; HERV-W; Temelimab; Post-COVID-19; PASC syndrome; Neuropsychiatric sequelae
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temelimab 54mg/kg (Experimental): Monthly IV repeated dose in addition to standard of care
  Interventions: Drug: Temelimab 54mg/kg
- Placebo (Placebo Comparator): Monthly IV repeated dose in addition to standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Temelimab 54mg/kg — Temelimab 54mg/kg will be given as monthly (every 4 weeks) intravenous (IV) infusion over 24 weeks (6 infusions in total)
  Arms: Temelimab 54mg/kg
Drug: Placebo — Placebo will be given as monthly (every 4 weeks) intravenous (IV) infusion over 24 weeks (6 infusions in total)
  Arms: Placebo

SUMMARY:
This study is a Phase 2, 24-week, randomized, prospective, double-blind, multicenter study in patients experiencing neuropsychiatric symptoms and functional impairment in the course of PASC. The purpose of the study is to evaluate the efficacy and safety of Temelimab as a treatment for PASC neuropsychiatric symptoms in patients who had severe acute respiratory syndrome coronavirus - type 2 (SARS-CoV-2) infection but did not undergo intensive care treatment during the acute period. Patients meeting eligibility criteria will be randomized to Temelimab or placebo in a 1:1 ratio via interactive voice/web response system to obtain 182 protocol completers. The randomization will be stratified by age (≤65 years versus >65 years).

ELIGIBILITY:
Main Inclusion Criteria:

* PASC Syndrome in accordance with NICE criteria with neuropsychiatric symptoms still occurring >12 weeks after their first appearance.
* Has had a SARS-CoV-2-positive diagnostic test (using a validated SARS-CoV-2 antigen, reverse transcription polymerase chain reaction [RT-PCR], or other molecular diagnostic assay, and an appropriate sample such as nasopharyngeal [NP], nasal, oropharyngeal [OP], or saliva). In case that the local standard of care did not foresee the previously mentioned tests, a confirmed SARS-CoV-2 nucleocapsid or membrane antibody test associated to a medical report documenting the date of COVID-19 clinical diagnostic, will be accepted.
* PROMIS Fatigue SF 7a total raw score ≥21 with onset of fatigue post coronavirus disease 2019 (COVID-19) infection.
* Patients affected with at least one of the following measures of objective impairment of cognitive function or of quality of life as defined by: i. Token Motor Test ≥1 z-score below the age/sex-adjusted mean ii. EQ5D-5L: Presence of at least 1 score ≥3 in any of the 5 variables of EQ5D-5L questionnaire (mobility; self-care; usual activities; pain/discomfort; anxiety/depression) iii. PQD-20 ≥27
* HERV-W ENV positive as defined by automated capillary western system, specific signal level over background noise (S/N) >1.

Main Exclusion Criteria:

* Intubation and mechanical ventilation in the course of COVID19 or reception of convalescent COVID19 plasma treatment at any time prior to study entry
* Major psychiatric conditions including but not restricted to (e.g. attention deficit/hyperactivity disorder, substance use disorder, schizophrenia documented in patient history or diagnosed using M.I.N.I), at the discretion of the site investigator, these do not refer to patients with typical mild to moderate symptoms of depression and anxiety associated with PASC
* Neurological signs and symptoms including change in level of consciousness, seizures, movement disorders or focal neurological deficits, disorders of the central nervous system with tissue damage or a pre-COVID-19 diagnosis of Chronic Fatigue Syndrome documented in the patient history or diagnosed during the neurological examination
* Current immunosuppressive//immunomodulating medication (e.g., azathioprine, tacrolimus, cyclosporine, methotrexate, hydroxychloroquine, cytotoxic chemotherapy, or neutralizing antibodies against SARS-CoV-2 epitopes) or therapy with HIV protease inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Improvement in fatigue in PASC patients | 24 weeks
  Occurrence of an improvement in fatigue, measured by a decrease of ≥3 points in the Patient-Reported Outcomes Measurement Information System Fatigue Short Form 7a (PROMIS Fatigue SF 7a) score, at Week 24 as compared to baseline.

SECONDARY OUTCOMES:
Fatigue | 24 weeks
  Change from baseline to Week 24 in the Severity of fatigue as measured by the PROMIS Fatigue SF 7a score
Cognitive function | 24 weeks
  Change from baseline to Week 24 in 5 domain scores (verbal memory test, digit sequencing test, Token Motor Test, verbal semantic and letter fluency, and Tower of London) as measured by BAC tests
Cognitive function | 24 weeks
  Change from baseline to Week 24 in Symbol Digit Modalities Test (SDMT) score
Cognitive function | 24 weeks
  Change from baseline to Week 24 in Cognitive function as measured by the composite score of the BAC excluding symbol coding test
Cognitive function | 24 weeks
  Change from baseline to Week 24 in Cognitive function as measured by the Perceived Deficits Questionnaire, 20 items (PDQ-20)
Anxiety | 24 weeks
  Change from baseline to Week 24 in Severity of anxiety as measured by the Generalized Anxiety Disorder, 7 Items (GAD 7)
Depression | 24 weeks
  Change from baseline to Week 24 in Severity of depression as measured by the Patient Health Questionnaire, 9 Items (PHQ-9)
Overall quality of Life | 24 weeks
  Change from baseline to Week 24 in Overall quality of life as measured by the European Quality of Life 5 Dimensions, 5 Levels (EQ5D-5L)
Functional impairment | 24 weeks
  Change from baseline to Week 24 in Level of functional impairment as measured by the Sheehan Disability Scale (SDS)
Post-COVID-19 Functional Status | 24 weeks
  Change from baseline to Week 24 in Post-COVID-19 Functional Status Scale (PCFS)
Safety and tolerability of Temelimab in PASC patients | 24 weeks
  Incidence of serious AEs [SAEs], AEs and analysis of physical examination findings, clinical laboratory values results

CONTACTS AND LOCATIONS:
Overall Officials: David LEPPERT, MD, Study Director — GeNeuro SA
Locations (14):
- Italy (4):
  - Clinica Metabolica dell'Università di Modena e Reggio Emilia, Modena
  - U.O.C. Malattie Infettive Tor Vergata, Policlincio Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Hospital of Vipiteno, Sterzing
- Spain (5):
  - Ace Alzheimer Center, Barcelona
  - Private clinic Blue Healthcare, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital General Universitario- Servicio de Medicina Interna, Valencia
  - Hospital Royo Villanova, Zaragoza
- Switzerland (5):
  - REHAB Clinic for Neurorehabilitation and Paraplegiology, Basel
  - Inselspital Bern University Hospital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Geneva University Hospital, Geneva
  - Centre hospitalier du Valais Romand (CHVR) - Hôpital du Valais, Sion